CLINICAL TRIAL: NCT02207322
Title: Randomized Study of a Targeted Inpatient Supportive Care Intervention in Patients Hospitalized for Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: Supportive Care Intervention In Patients Hospitalized For Hematopoietic Stem Cell Transplantation (Shield)
Acronym: SHIELD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, El-Jawahri, Areej,M.D., Director MGH BMT Survivorship Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-241
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Results first posted 2019-03-06 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Complication of Transplant
Keywords: Hematopoietic stem cell transplantation (HSCT); autologous stem cell transplant; allogeneic stem cell transplant
MeSH Terms: interventions — Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard transplant care (No Intervention): * Patient Enrollment and Caregiver Enrollment (within 72 hours of hospital)
    -- Complete baseline data collection, and registration
  * Patient Randomization
  * Standard transplant oncology care
    -- Palliative care consults only upon request
  * Longitudinal Data Collection (patient & family caregivers)
    * Week-2 of hospitalization
    * 3-months, and 6-months post HSCT
- transplant with early palliative care (Experimental): * Standard transplant oncology care with early palliative care
  * Patient Enrollment and Caregiver Enrollment (within 72 hours of patient enrollment)
    --Complete baseline data collection, and registration Intervention description: Inpatient palliative care intervention description: 1st visit within 72 hours of randomization, At least twice weekly follow up visits
  * Longitudinal Data Collection (patient & family caregivers)
    * Week-2 of hospitalization
    * 3-months, and 6-months post HSCT
  Interventions: Other: transplant with early palliative care

INTERVENTIONS:
Other: transplant with early palliative care — the intervention include integrating early palliative care with standard transplant care to evaluate and treat patients' symptoms during stem cell transplantation
  Arms: transplant with early palliative care

SUMMARY:
The main purpose of this study is to assess whether early integration of palliative and supportive care services in care of patients hospitalized for hematopoietic stem cell transplantation (HSCT) can improve patients' and family caregivers' quality of life and mood.

DETAILED DESCRIPTION:
This research study is evaluating the impact of early involvement of supportive care team working with the transplant oncology team will have on the quality of life, symptoms, and mood of patients undergoing stem cell transplantation.

The purpose of this research study is to find out whether introducing patients and families undergoing stem cell transplantation to the palliative care team that specializes in symptom management can improve the physical and psychological symptoms that patients and families experience during hospitalization for stem cell transplantation.

The study will use a series of questionnaires to measure participant's and their caregivers' quality of life, physical symptoms, and mood. Study questionnaires will be completed in the hospital or clinic with assistance provided as needed

ELIGIBILITY:
Inclusion Criteria:

* Patients Eligibility Criteria:

  * Adult patients (≥18 years) with hematologic malignancy admitted to Massachusetts General Hospital for HSCT are eligible for the study.
  * Ability to speak English or able to complete questionnaires with minimal assistance required from an interpreter or family member.
* Caregivers Eligibility Criteria:

  * Adult caregivers (>18 years) of patients undergoing HSCT at MGH who agreed to participate in study.
  * A relative or a friend, identified by the patient who either lives with the patient or has in-person contact with him or her at least twice per week.
  * Ability to read questions in English or willing to complete questionnaires with the assistance of an interpreter.

Exclusion Criteria:

* Patients with prior history of HSCT.
* Patients undergoing HSCT for a benign hematologic condition (myelodysplastic syndrome (MDS) is not considered a benign hematologic condition and patients with MDS are eligible for the study)
* Significant uncontrolled psychiatric disorder (psychotic disorder, bipolar disorder, major depression) or other co-morbid disease (dementia, cognitive impairment), which the treating clinician believes prohibits informed consent or participation in the study.
* Patients enrolled on other supportive care intervention trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Areej El-Jawahri, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Newcomb R, Amonoo HL, Kavanaugh AR, Wharton KC, Rowland M, Fausto J, Webb J, Jackson V, Greer JA, Temel JS, Lark P, Rabideau DJ, O'Brien K, LeBlanc TW, Lee SJ, El-Jawahri A. Factors associated with early quality-of-life response to palliative care during hematopoietic cell transplantation. Blood Adv. 2025 May 13;9(9):2033-2043. doi: 10.1182/bloodadvances.2024014574. PMID 39908568
- [Derived] El-Jawahri A, LeBlanc T, VanDusen H, Traeger L, Greer JA, Pirl WF, Jackson VA, Telles J, Rhodes A, Spitzer TR, McAfee S, Chen YA, Lee SS, Temel JS. Effect of Inpatient Palliative Care on Quality of Life 2 Weeks After Hematopoietic Stem Cell Transplantation: A Randomized Clinical Trial. JAMA. 2016 Nov 22;316(20):2094-2103. doi: 10.1001/jama.2016.16786. PMID 27893130

RESULTS

PARTICIPANT FLOW:
Groups:
- Transplant With Early Palliative Care: * Standard transplant oncology care with early palliative care
  * Patient Enrollment and Caregiver Enrollment (within 72 hours of patient enrollment)
    --Complete baseline data collection, and registration Intervention description: Inpatient palliative care intervention description: 1st visit within 72 hours of randomization, At least twice weekly follow up visits
  * Longitudinal Data Collection (patient & family caregivers)
    * Week-2 of hospitalization
    * 3-months, and 6-months post HSCT
  transplant with early palliative care: the intervention include integrating early palliative care with standard transplant care to evaluate and treat patients' symptoms during stem cell transplantation
Period: Overall Study
Arm/Group | Standard Transplant Care | Transplant With Early Palliative Care
Started | 79 | 81
Week-2 | 77 | 80
3-month | 74 | 75
Completed (6-month) | 70 (6-month) | 71 (6-month)
Not Completed | 9 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Transplant Care | Transplant With Early Palliative Care | Total
Number analyzed (Participants) | 79 | 81 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (14.1) | 57.2 (12.7) | 57.1 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 48 | 91
  Male | 36 | 33 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 78 | 78 | 156
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Functional Assessment of Cancer Therapy - Bone Marrow Transplant (FACT-BMT) Score at Week-2
Description: Compare quality of life (QOL) (FACT-BMT) scores at week-2 (day+5 for autologous, day +8 for myeloablative or reduced intensity allogeneic HSCT) adjusting for baseline QOL scores between the study arms. Score range 0-164 with higher scores indicating better quality of life
Time Frame: week-2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Transplant Care | Transplant With Early Palliative Care
Number analyzed (Participants) | 77 | 80
units on a scale | 86.60 [82 to 91.20] | 94.33 [89.81 to 98.84]

2. Secondary Outcome: FACT-BMT Score at 3 Months
Description: adjusted patient-reported quality of life (QOL) at 3-month adjusting for baseline QOL scores Score range 0-164 with higher scores indicating better quality of life
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Transplant Care | Transplant With Early Palliative Care
Number analyzed (Participants) | 74 | 75
units on a scale | 106.66 [102.91 to 110.41] | 112.00 [108.28 to 115.73]

3. Secondary Outcome: FACT-BMT Score at 6 Months
Description: compare quality of life between the two study arms at 6 months adjusting for baseline scores Score range 0-164 with higher scores indicating better quality of life
Time Frame: 6 Months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Transplant Care | Transplant With Early Palliative Care
Number analyzed (Participants) | 70 | 71
units on a scale | 109.39 [105.38 to 113.41] | 112.11 [108.12 to 116.10]

4. Secondary Outcome: Depression Symptoms at Week-2 Using the Hospital Anxiety and Depression Scale (HADS)
Description: compare depression symptoms using HADS at week-2 adjusting for baseline scores HADS-depression scale range 0-21 with higher score indicating higher depression symptoms
Time Frame: week-2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Transplant Care | Transplant With Early Palliative Care
Number analyzed (Participants) | 77 | 80
units on a scale | 8.49 [7.59 to 9.39] | 6.74 [5.86 to 7.63]

5. Secondary Outcome: Depression Symptoms at 3 Month Using the Hospital Anxiety and Depression Scale (HADS)
Description: compare depression symptoms using HADS at 3 months adjusting for baseline scores HADS-depression scale range 0-21 with higher score indicating higher depression symptoms
Time Frame: 3 month
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Transplant Care | Transplant With Early Palliative Care
Number analyzed (Participants) | 74 | 74
units on a scale | 5.19 [4.45 to 5.93] | 3.49 [2.75 to 4.23]

6. Secondary Outcome: Depression Symptoms at 6 Month Using the Hospital Anxiety and Depression Scale (HADS)
Description: Compare depression symptoms using HADS at 6 months adjusting for baseline scores HADS-depression scale range 0-21 with higher score indicating higher depression symptoms
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Transplant Care | Transplant With Early Palliative Care
Number analyzed (Participants) | 70 | 71
units on a scale | 4.66 [3.93 to 5.38] | 3.45 [2.70 to 4.19]

7. Secondary Outcome: Anxiety Symptoms at Week-2 Using the Hospital Anxiety and Depression Scale (HADS)
Description: compare anxiety symptoms using HADS at week-2 adjusting for baseline scores HADS-anxiety scale range 0-21 with higher score indicating higher anxiety symptoms
Time Frame: week-2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Transplant Care | Transplant With Early Palliative Care
Number analyzed (Participants) | 77 | 80
units on a scale | 6.33 [5.64 to 7.02] | 4.08 [3.40 to 4.75]

8. Secondary Outcome: Anxiety Symptoms at 3 Months Using the Hospital Anxiety and Depression Scale (HADS)
Description: compare anxiety symptoms using HADS at 3 months adjusting for baseline scores HADS-anxiety scale range 0-21 with higher score indicating higher anxiety symptoms
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Transplant Care | Transplant With Early Palliative Care
Number analyzed (Participants) | 74 | 74
units on a scale | 4.84 [4.15 to 5.53] | 4.08 [3.39 to 4.78]

9. Secondary Outcome: Anxiety Symptoms at 6 Months Using the Hospital Anxiety and Depression Scale (HADS)
Description: compare anxiety symptoms using HADS at 6 months adjusting for baseline scores HADS-anxiety scale range 0-21 with higher score indicating higher anxiety symptoms
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Transplant Care | Transplant With Early Palliative Care
Number analyzed (Participants) | 72 | 69
units on a scale | 4.74 [3.99 to 5.49] | 4.13 [3.36 to 4.90]

10. Secondary Outcome: Depression Scores Using Patient Health Questionnaire-9 (PHQ9) at Week-2
Description: compare PHQ-9 score at week-2 between study arms adjusting for baseline scores the PHQ-9 range from 0-27 with higher scores indicating higher depression
Time Frame: week 2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Transplant Care | Transplant With Early Palliative Care
Number analyzed (Participants) | 77 | 80
units on a scale | 9.52 [8.42 to 10.63] | 8.25 [7.16 to 9.33]

11. Secondary Outcome: Depression Scores Using Patient Health Questionnaire-9 (PHQ9) at 3 Months
Description: compare PHQ-9 score at 3-months between study arms adjusting for baseline scores the PHQ-9 range from 0-27 with higher scores indicating higher depression
Time Frame: 3-month
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Transplant Care | Transplant With Early Palliative Care
Number analyzed (Participants) | 74 | 75
units on a scale | 5.94 [5.02 to 6.86] | 3.82 [2.91 to 7.47]

12. Secondary Outcome: Depression Scores Using Patient Health Questionnaire-9 (PHQ9) at 6 Months
Description: compare PHQ-9 score at 6-months between study arms adjusting for baseline scores the PHQ-9 range from 0-27 with higher scores indicating higher depression
Time Frame: 6-month
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Transplant Care | Transplant With Early Palliative Care
Number analyzed (Participants) | 71 | 71
units on a scale | 5.58 [4.57 to 6.60] | 3.95 [2.93 to 4.98]

13. Secondary Outcome: Fatigue Scores (as Measured by FACT-Fatigue) at Week-2
Description: examine change in fatigue scores at week-2 adjusting for baseline scores Fatigue score ranges from 0 to 52 with higher scores indicating lower fatigue symptoms
Time Frame: week-2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Transplant Care | Transplant With Early Palliative Care
Number analyzed (Participants) | 77 | 79
units on a scale | 23.71 [21.11 to 26.31] | 27.59 [25.01 to 30.16]

14. Secondary Outcome: Fatigue Scores (as Measured by FACT-Fatigue) at 3 Months
Description: compare change in fatigue scores at 3 months adjusting for baseline scores Fatigue score ranges from 0 to 52 with higher scores indicating lower fatigue symptoms
Time Frame: 3-months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Transplant Care | Transplant With Early Palliative Care
Number analyzed (Participants) | 74 | 73
units on a scale | 35.60 [33.43 to 37.77] | 37.60 [35.42 to 39.79]

15. Secondary Outcome: Symptom Burden (as Measured by the Edmonton Symptom Assessment Scale) at Week-2
Description: compare symptom burden as measured by Edmonton Symptom Assessment Scale at week-2 adjusting for baseline scores Symptoms burden range is from 0-90 with higher scores indicating higher symptom burden
Time Frame: week-2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Transplant Care | Transplant With Early Palliative Care
Number analyzed (Participants) | 77 | 75
units on a scale | 37.74 [34.09 to 41.40] | 31.49 [27.79 to 35.19]

16. Secondary Outcome: Patient-reported Post-Traumatic Stress Disorder (PTSD) as Measured by the PTSD Checklist at 3 Months
Description: Compare patient-reported Post-Traumatic Stress Disorder (PTSD) as measured by the PTSD checklist at 3 months PTSD score ranges from 17-85 with higher scores indicating higher PTSD symptoms
Time Frame: 3-months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Transplant Care | Transplant With Early Palliative Care
Number analyzed (Participants) | 67 | 72
units on a scale | 25.79 [23.79 to 27.79] | 21.44 [19.53 to 23.35]

17. Secondary Outcome: Patient-reported Post-Traumatic Stress Disorder (PTSD) as Measured by the PTSD Checklist at 6 Months
Description: Compare patient-reported Post-Traumatic Stress Disorder (PTSD) as measured by the PTSD checklist at 6 months PTSD score ranges from 17-85 with higher scores indicating higher PTSD symptoms
Time Frame: 6-months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Transplant Care | Transplant With Early Palliative Care
Number analyzed (Participants) | 71 | 68
units on a scale | 26.18 [23.96 to 28.39] | 22.15 [19.91 to 24.40]

18. Other Pre Specified Outcome: Caregiver Quality of Life
Description: we will use the CareGiver Oncology QOL questionnaire (CarGOQOL) to compare caregiver QOL at week-2 between the study arms caregiver quality of life score ranges from 0-120 with higher scores indicating better caregiver quality of life
Time Frame: week-2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Transplant Care | Transplant With Early Palliative Care
Number analyzed (Participants) | 40 | 46
units on a scale | 113.32 [107.79 to 118.85] | 118.71 [114.40 to 123.03]

19. Other Pre Specified Outcome: Caregiver Depression Symptoms Using Hospital Anxiety and Depression Scale (HADS)
Description: compare caregiver depression at week-2 using hospital anxiety and depression scale (HADS) caregiver depression score ranges from 0-21 with higher score indicating higher depression symptoms
Time Frame: week 2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Transplant Care | Transplant With Early Palliative Care
Number analyzed (Participants) | 42 | 46
units on a scale | 6 [4.51 to 7.49] | 4.05 [3.01 to 5.10]

20. Other Pre Specified Outcome: Caregiver Anxiety Symptoms Using Hospital Anxiety and Depression Scale (HADS)
Description: compare caregiver anxiety at week-2 using hospital anxiety and depression scale (HADS)
Time Frame: week 2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Transplant Care | Transplant With Early Palliative Care
Number analyzed (Participants) | 42 | 46
units on a scale | 6.54 [5.09 to 7.99] | 6.24 [5.10 to 7.37]

ADVERSE EVENTS:
Time Frame: 1 year
Description: this is a supportive care trial. there are no adverse events that have been observed
Arm/Group | Standard Transplant Care | Transplant With Early Palliative Care
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/81
Other Adverse Events (participants affected / at risk) | 0/79 | 0/81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No